CLINICAL TRIAL: NCT06391775
Title: First-In-Human, Open-Label, Dose Escalation Trial With Expansion Cohorts to Evaluate the Safety and Preliminary Efficacy of GEN1055 as Monotherapy and as Combination Therapy in Subjects With Malignant Solid Tumors
Brief Title: Trial to Assess the Safety and Preliminary Efficacy of GEN1055 on Malignant Solid Tumors as Monotherapy and as Combination Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to strategic decision
Sponsor: Genmab (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1055-01; 2023-507049-28-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Malignant Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): GEN1055 will be administered as monotherapy and in combination with a fixed dose of pembrolizumab.
  Interventions: Biological: GEN1055; Biological: Pembrolizumab
- Expansion (Experimental): GEN1055 will be administered as monotherapy or in combination with pembrolizumab or in combination with pembrolizumab and standard chemotherapy in separate expansion cohorts, at a dose level selected from the Dose Escalation part.
  Interventions: Biological: GEN1055; Biological: Pembrolizumab; Drug: Standard Chemotherapy

INTERVENTIONS:
Biological: GEN1055 — Intravenous (IV) administration.
Biological: Pembrolizumab — IV administration
Drug: Standard Chemotherapy — IV administration
  Arms: Expansion

SUMMARY:
The goal of this trial is to learn about the antibody GEN1055 when it is used alone and when it is used together with another antibody cancer drug, pembrolizumab (with or without chemotherapy), for treatment of participants with certain types of cancer. Participants will receive either GEN1055 alone, GEN1055 with pembrolizumab, or GEN1055 with pembrolizumab and chemotherapy. All participants will receive active drug; no one will receive placebo.

This trial has 2 parts. The purpose of the first part is to find out if GEN1055 is safe and to find out the doses of GEN1055 to use alone and to use with pembrolizumab. The purpose of the second part is to give GEN1055 to more participants to see how well the doses of GEN1055 that were selected in the first part work against cancer alone and how well they work with pembrolizumab (with or without other chemotherapy).

A participant will receive trial treatment up to a maximum of 24 months for pembrolizumab-containing regimens, or until:

* the cancer progresses.
* there are side effects requiring that treatment be stopped.
* the participant decides to not participate further in this trial.
* the doctor believes it is in the participant's best interest to stop treatment.

Participation in the trial will require visits to the site. For the first 12 weeks there will be weekly visits and after that, visits will be every 3 weeks. At site visits, there will be various tests (such as blood draws) and procedures (such as recording of heart activity, computed tomography (CT) scans) to monitor whether the treatment is safe and effective. The trial duration (including screening, treatment, and follow-up) for each participant will be about 39 months.

DETAILED DESCRIPTION:
This is a multi-center trial and will be conducted in two parts: dose escalation (phase 1a/1b) and expansion (phase 2a).

The Dose Escalation part of the trial will evaluate dose-limiting toxicities (DLTs) to determine the recommended phase 2 dose (RP2D), and if reached, the maximum tolerated dose (MTD) in participants with locally advanced or metastatic solid tumors.

The Expansion part will evaluate safety, tolerability, mechanism of action (MoA), immunogenicity, pharmacokinetic (PK), and initial antitumor activity of the selected doses and schedules in selected tumor indications.

ELIGIBILITY:
Inclusion Criteria:

All cohorts:

* Be at least 18 years of age.
* Have measurable disease according to RECIST v1.1.
* Provide all pre-baseline scans since failure of last prior therapy (ie, documented radiographic progressive disease [PD]), if available.
* Have Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 to 1 at screening and on C1D1 pretreatment.
* Provide a biopsy (ie, formalin-fixed paraffin-embedded slides/block). A fresh biopsy taken during the screening period is preferred, unless medically unfeasible and after review and approval by the sponsor. If this cannot be provided, a biopsy taken after failure/stop of last prior treatment and taken within 6 months prior to C1D1 may be provided.

Phase 1a and 1b- Dose Escalation:

* Have histologically or cytologically confirmed non-Central Nervous System (CNS) primary solid tumors who have metastatic or advanced disease.
* Have progressed on standard of care (SoC) therapy which should include platinum-based chemotherapy and anti-PD/PD-L1 therapies, if applicable for the tumor type, or for whom there is no available standard therapy likely to provide clinical benefit, and for whom experimental therapy with GEN1055 or GEN1055+pembrolizumab may be beneficial, in the opinion of the investigator.

Phase 2a - Expansion:

Inclusion criteria specific to selected tumor indications may apply.

Exclusion Criteria:

* Has uncontrolled intercurrent illness, including but not limited to:

  * Ongoing or active infection requiring IV treatment with anti-infective therapy administered less than 2 weeks prior to first dose (including coronavirus disease 2019 [COVID-19] infection).
  * Significant cardiovascular impairment including:

    i) Symptomatic congestive heart failure (Class III or IV as classified by the New York Heart Association), unstable angina pectoris, or cardiac arrhythmia.

ii) Uncontrolled hypertension defined as systolic blood pressure ≥160-millimeter (mm) Hg and/or diastolic blood pressure ≥100 mm Hg, despite optimal medical management.

iii) Prolonged corrected QT interval at baseline of ≥470 milliseconds using Fridericia's QT correction formula.

* Ongoing or recent (within 1 year of screening) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs).
* History of grade 3 or higher irAEs that led to treatment discontinuation of a checkpoint inhibitor (CPI). A participant with irAEs below grade 3 that led to discontinuation should be discussed with the sponsor. Grade 3 irAEs that have fully recovered may also be discussed.
* History of chronic liver disease (eg, alcoholic hepatitis or nonalcoholic steatohepatitis), drug-related or autoimmune hepatitis, or evidence of hepatic cirrhosis.
* Evidence of interstitial lung disease.
* Ongoing pneumonitis (any grade) including any radiological change of ongoing pneumonitis at baseline or history of noninfectious drug-, immune-, or radiation-related pneumonitis that has required steroids.

  * Has been exposed to any of the following prior therapies/treatments within the specified timeframes:
* Treatment with an anticancer agent within 4 weeks or for systemic therapies within 5 half-lives of the drug, whichever is shorter, prior to trial treatment administration.
* Condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first treatment. Inhaled or topical steroids, and adrenal or pituitary replacement steroid >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Has received granulocyte or granulocyte/macrophage colony-stimulating factor support within 2 weeks prior to first trial treatment administration or is chronically transfusion-dependent.
* RT within 14 days before the planned first dose of trial treatment. Palliative RT of bone metastases up to 7 days prior to C1D1 will be allowed.

  * Hepatitis (testing for hepatitis B or C is not required unless mandated by local health authority):
* Hepatitis B virus (HBV): Has a medical history or positive serology for HBV (defined as positive for hepatitis B surface antigen or HBV deoxyribonucleic acid [DNA]).

  i) Above is not exclusionary if deemed due to vaccination, resolved natural infection, or passive immunization due to immunoglobulin therapy.
* Hepatitis C virus (HCV): Known active HCV infection (defined as positive for HCV ribonucleic acid [RNA] [qualitative]).

Note: Other protocol defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Number of Participants With Adverse Events (AEs) | From first dose date up to end of the survival follow up period (up to 39 months)
Dose Escalation: Number of Participants With DLTs | During first cycle (21 days) for each cohort
  Toxicities will be graded for severity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0.
Expansion: Overall Response Rate (ORR) | Up to 39 months
  ORR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 as assessed by investigator.

SECONDARY OUTCOMES:
Dose Escalation and Expansion: Maximum (peak) Plasma Concentration (Cmax) of GEN1055 | Predose and postdose at multiple timepoints of each Cycle up to end of treatment (Cycle length=21 days)
Dose Escalation and Expansion: Time to Reach Cmax (Tmax) for GEN1055 | Predose and postdose at multiple timepoints of each Cycle up to end of treatment (Cycle length=21 days)
Dose Escalation and Expansion: Plasma Trough (Pre-dose) Concentrations (Ctrough) of GEN1055 | Predose and postdose at multiple timepoints of each Cycle up to end of treatment (Cycle length=21 days)
Dose Escalation and Expansion: Area Under the Concentration-Time Curve from Time 0 to Last Quantifiable Sample (AUC0-tlast) for GEN1055 | Predose and postdose at multiple timepoints of each Cycle up to end of treatment (Cycle length=21 days)
Dose Escalation and Expansion: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-inf) for GEN1055 | Predose and postdose at multiple timepoints of each Cycle up to end of treatment (Cycle length=21 days)
Dose Escalation and Expansion: Half-life (t½) of GEN1055 | Predose and postdose at multiple timepoints of each Cycle up to end of treatment (Cycle length=21 days)
Dose Escalation and Expansion: Clearance (CL) of GEN1055 From the Plasma | Predose and postdose at multiple timepoints of each Cycle up to end of treatment (Cycle length=21 days)
Dose Escalation and Expansion: Number of Participants with Anti-Drug Antibody (ADA) | Predose and postdose at multiple timepoints of each Cycle up to end of treatment (Cycle length=21 days)
  Serum samples will be screened for ADAs binding to GEN1055 and the titer of confirmed positive samples will be reported.
Dose Escalation: ORR | Up to 39 months
  ORR is defined as the proportion of participants with BOR of CR or PR according to RECIST v1.1 as assessed by investigator.
Dose Escalation and Expansion: Duration of Response (DOR) | Up to 39 months
  DOR based on investigator assessment is defined as the time from the first documentation of response (CR or PR) to the date of Progressive Disease (PD) or death, whichever occurs earlier according to RECIST v1.1 as assessed by investigator.
Dose Escalation and Expansion: Time to Response (TTR) | Up to 39 months
  TTR based on investigator assessment is defined as the time from Cycle 1 Day 1 (C1D1) to first documentation of objective response (CR or PR) in participants achieving PR or CR according to RECIST v1.1 as assessed by investigator.
Dose Escalation and Expansion: Disease Control Rate (DCR) | Up to 39 months
  The DCR is defined as the proportion of participants with BOR of CR, PR, or Stable Disease (SD) according to RECIST v1.1 as assessed by investigator.
Expansion: Overall Survival (OS) | Up to 39 months
  OS is defined as the time from C1D1 to the date of death due to any cause.
Expansion: Progression Free Survival (PFS) | Up to 39 months
  PFS is defined as the time from C1D1 to first documented PD or death due to any cause, whichever occurs earlier according to RECIST v1.1 as assessed by investigator.
Expansion: Number of Participants With AEs | From first dose date up to end of the survival follow up period (up to 39 months)

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (4):
- Yale-New Haven Hospital, New Haven, Connecticut, United States
- Spain (3):
  - Hospital Universtari Val D´Hebron, Barcelona
  - Start Madrid Ciocc Hm Sanchinarro, Madrid
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No